CLINICAL TRIAL: NCT05039294
Title: The Effect Of A School-Based Physical Activity Educational Program On Adolescents' Physical Activity-related Knowledge, Performance, And Self-Efficacy
Brief Title: The Effect Of A School-Based Physical Activity Educational Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Nahla Ali, Associate professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20200023
Record Dates: First submitted 2021-08-12; First posted 2021-09-09 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Improve Physical Activity
Keywords: physical activity; self-efficacy; school programs; educational program
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: using code number and randomly assigned to intervention and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): provided the educational programs with all contents, and follow up after one month
  Interventions: Behavioral: School-Based Physical Activity Educational Program
- control (No Intervention): received no intervention, but assessed pre-post

INTERVENTIONS:
Behavioral: School-Based Physical Activity Educational Program — The structure of the educational sessions includes physical education lectures, group discussions, videos, training sessions, physical activities diaries, short quizzes, and feedback after each session. The educational programs were conducted among students with intervention groups at two-level individually and in school. The individual-level includes classroom lectures that mainly emphasized the health benefits of physical activity and provided necessary information about physical activity fitness for 60 minutes and were given weekly for four weeks. In coordination with the school sports teacher, training sessions included moderate to vigorous physical activities for 45 minutes twice weekly for four weeks
  Arms: intervention

SUMMARY:
Regular physical activity of different intensity has many significant benefits for all ages, particularly adolescents. School-based educational programs about physical activity were found to increase the level of physical activity among adolescents positively. However, among adolescents in Jordan, few studies measured the impact of school-based educational programs on students' physical activity and knowledge levels. There is no single study that measured the students' physical activity self-efficacy. The study aimed to assess the effectiveness of a school-based physical activity program on adolescents' knowledge of the physical activity, physical performance, and physical self-efficacy. A Randomized Control trial (RCT) design was used among 210 8th grade school students (boys and girls) from four governmental schools in North of Jordan .

DETAILED DESCRIPTION:
Background: Regular physical activity of different intensity has many significant benefits on the health of all ages, particularly adolescents. School-based educational programs about physical activity were found to increase the level of physical activity among adolescents positively. However, among adolescents in Jordan, few studies measured the impact of school-based educational programs on students' level of physical activity and knowledge, and there is no single study that measured the students' physical activity self-efficacy.

Aim: To assess the effectiveness of a school-based physical activity program on adolescents' knowledge of physical activity, physical performance, and physical self-efficacy.

Methods: A Randomized Control trial (RCT) design was used among 210 8th grade school students (boys and girls) from four governmental schools in North of Jordan during December and January. Physical Activity Questionnaire for older children (PAQ-C) scales, Physical self-efficacy scale, and Knowledge of Physical Activity scale were used to collect students' data. The duration of the educational program was four weeks, with a total of 7 hours. Ethical approval was approached from the Committee on Human Subjects Research at Jordan University of Science and Technology and the Ministry of Education before the data collection.

ELIGIBILITY:
Inclusion Criteria:

* all students boys and girls in 8th grade from selected schools affiliated with eight educational directorates of the Irbid governorate,
* who are ready to participate in the educational program and meet the inclusion criteria.

Exclusion Criteria:

* Students who have any medical problems (asthma, diabetes, cardiac problems) and physical disabilities were excluded.

Ages: 13 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Boys and girls are eligible
Enrollment: 210 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Knowledge | baseline pre-intervention, and immediately after the intervention
  Adolescents' Physical Activity-Related Knowledge: This section was developed by the researcher based on previous literature. The questionnaire contained eighteen questions to assess student knowledge about the definition of physical activity, exercise, health, and physical fitness. Types of physical activity, physical activity benefits, and negative consequences of physical inactivity on health, and recommendation. Each of the eighteen items has three alternatives: true, false, and do not know. The total knowledge score was used based on the percentages of the correctly answered questions.
physical activity level | baseline pre-intervention, and immediately after the intervention
  Physical activity performance: Physical Activity Questionnaires for older children (PAQ-C) is used to assess moderate to vigorous physical activity levels over the past 7 days (Crocker et al.,1997). It includes eight questions, each one scored on 5 point scale. Item 1 (Spare time activity) takes the mean of all activities ("no" activity being a 1, "7 times or more" being a 5) on the activity checklist to form a composite score for item 1. Items 2 to 8 (PE, recess, lunch, right after school, evening, weekends, and describes you best), the answers reflect the level of physical activity for each item from lowest activity response to the highest activity response. Then used the reported value is determined for each item (the lowest activity response being a 1 and the highest activity response being a 5). Item 9 reflects the mean of physical activity during the week ("none" being a 1, "very often" being a 5) to form a composite score for item 9
self-efficacy | baseline pre-intervention, and immediately after the intervention
  physical activity self-efficacy":The final validated modified version of the physical activity self-efficacy scale adolescent's protocol questionnaire (Motl et al., 2000) consists of 8 items used in this study to measure physical activity self-efficacy. The scale contains two sections: self-management and social support. Self-management of the physical activity section consists of 6 items related to cognitive and behavioral factors that may increase or decrease physical activity participation. Social support was measured by two items which are support from family and friends. The students were asked to choose from 5 items on a Likert scale. The scoring ranged from 1 (disagree a lot) to 5 (agree a lot). The total score of both sections ranged from 8- 40, higher scores indicate higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Nahla M. Al Ali, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Nahla M. Al Ali, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided